CLINICAL TRIAL: NCT06522672
Title: A Study to Assess the Effect of My Happy Flo on Alleviating Period Symptoms and Heavy Flows.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: My Happy Flo (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20436
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Menstrual Cramps; Women's Health; Fatigue
Keywords: Menstrual Health; Period Symptoms
MeSH Terms: conditions — Dysmenorrhea; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- My Happy Flo Supplement (Experimental): Participants will take two capsules of My Happy Flo daily, preferably in the morning with 8-10 oz of water and a meal, for three menstrual cycles.
  Interventions: Dietary Supplement: My Happy Flo

INTERVENTIONS:
Dietary Supplement: My Happy Flo — The intervention aims to alleviate period symptoms including heavy flows, prolonged periods, cramps, mood disturbances, energy levels, cycle regulation, and fatigue. Blood tests for Vitamin D and Iron levels will be conducted at Baseline and after the third menstrual cycle. Participants will complete validated questionnaires assessing period symptoms after each menstrual cycle.

SUMMARY:
This clinical study aims to evaluate the effectiveness of My Happy Flo, a dietary supplement, in alleviating period symptoms and heavy menstrual flows. The study involves 40 participants, who will take the supplement daily for three menstrual cycles. Primary outcomes, such as the severity of heavy flows, prolonged periods, cramps, mood, energy levels, cycle regulation, and fatigue, will be measured using validated questionnaires completed after each menstrual cycle. Secondary outcomes, including Vitamin D and Iron levels, will be assessed through blood tests at the beginning and end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 or over
* Experiencing heavy period flows
* Two or more self-reported symptoms (prolonged periods, cramps, poor mood, fatigue, irregular cycle)
* Signs of potential anemia or iron deficiency
* No known allergies to the product ingredients
* Willing to comply with study requirements and limit caffeine intake
* Generally healthy - do not live with any uncontrolled chronic disease

Exclusion Criteria:

* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
* A diagnosis of sports anemia within the previous 6 months
* Anyone with known severe allergic reactions that require an Epi-Pen
* Women who are pregnant, breastfeeding, or trying to conceive
* Anyone unwilling to follow the study protocol
* Anyone who has undergone any surgeries or invasive treatments (such as immunotherapy, chemotherapy, radiation, or biological cancer) in the last 30 days or has any planned for the next 12 weeks
* Anyone with a history of substance abuse
* Anyone currently participating or planning to participate in a research study
* Anyone taking prescription anticonvulsants (anti-seizure medications)
* Anyone taking prescription anticoagulant medications (blood thinners)
* Anyone taking any hormone-modulating medications (e.g., hormonal birth control, hormone replacement therapy, testosterone, tamoxifen, thyroid medications, etc.)
* History of hysterectomy, oophorectomy, or other surgery to the reproductive organs
* History of gynecologic cancer, such as cervical, ovarian, uterine, vaginal, or vulvar cancer
* Currently experiencing menopausal or perimenopausal symptoms
* Changes or cessation of hormonal birth control in the last three months
* Active or abnormal uterine/vaginal bleeding
* Resides in RI, NY, NJ, or AZ

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Improvement in Period Symptoms | Baseline (Day 0), Cycle 1, Cycle 2, and Cycle 3 - each Cycle is 28 days
  Measurement of heavy flows, prolonged periods, cramps, mood disturbances, energy levels, cycle regulation, and fatigue using validated questionnaires.

SECONDARY OUTCOMES:
Changes in Vitamin D Level | Baseline and Cycle 3 - each Cycle is 28 days
  Assessment of Vitamin D level through blood tests.
Changes in Iron Level | Baseline and Cycle 3 - each Cycle is 28 days
  Assessment of Iron level through blood tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No